CLINICAL TRIAL: NCT03628521
Title: Anlotinib-based Combination as First-line Treatment in Advanced Non-small Cell Lung Cancer: a Single Center, Three Arms and Exploratory Study
Brief Title: First-line Combination Treatment Based on Anlotinib
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Baohui Han, professor, Shanghai Chest Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTION
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer; Advanced Stage
Keywords: lung cancer; first-line; combination
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- arm A (Other): Anlotinib combined with erlotinib. Anlotinib will be given at a dose of 10mg once daily on days 1-14 of a 21-day cycle. Erlotinib will be given at a dose of 150mg once daily.
  Interventions: Drug: Anlotinib，Erlotinib，IBI308，Pemetrexed，gemcitabine，carboplatin
- arm B (Other): Anlotinib combined with chemotherapy. Anlotinib will be given at a dose of 12mg once daily on days 1-14 of a 21-day cycle. Pemetrexed (just for adenocarcinoma) will be given intravenously at a dose of 500mg per square meter of body surface area every 3 weeks; gemcitabine (just for squamous carcinoma) will be given intravenously at a dose of 1000mg per square meter of body surface area every 3 weeks; carboplatin will be given intravenously with a target area under the curve of 5 mg per milliliter per minute every 3 weeks.
  Interventions: Drug: Anlotinib，Erlotinib，IBI308，Pemetrexed，gemcitabine，carboplatin
- arm C (Other): Anlotinib combined with IBI308. Anlotinib will be given at a dose of 12mg once daily on days 1-14 of a 21-day cycle. IBI308 will be given intravenously at a dose of 200mg every 3 weeks.
  Interventions: Drug: Anlotinib，Erlotinib，IBI308，Pemetrexed，gemcitabine，carboplatin

INTERVENTIONS:
Drug: Anlotinib，Erlotinib，IBI308，Pemetrexed，gemcitabine，carboplatin — Patient harboring EGFR mutation will be enrolled into arm A. Patients without sensitive EGFR mutation will be assigned to either arm B or arm C based on patients' or treating physicians'choice

SUMMARY:
The aim of this study is to explore safety and therapeutic efficacy of anlotinib combined with erlotinib/chemotherapy/IBI308 as first-line treatment in advanced NSCLC patients. The primary endpoints of the study are safety and objective response rate (ORR);the secondary endpoints are disease control rate (DCR), progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients have voluntarily to join the study and give written informed consent for the study
2. Histologically documented, unresectable, inoperable, locally advanced, recurrent or metastatic stage IIIB or IV Non-Small Cell Lung Cancer (NSCLC)
3. A cytologic diagnosis is acceptable (i.e., FNA or pleural fluid cytology)
4. Mutation status including EGFR, ALK ROS are explicit;
5. At least 1 unidimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumours (RECIST) criteria.
6. Patients did not receive systemic anti-cancer therapy previously, including traditional Chinese medicine.
7. Able to comply with study and follow-up procedures
8. Age ≥ 18 years and ≤ 75, ECOG PS: 0~1, estimated survival duration more than 3 months;enough organ function;

8)Major organ function

1. For regular test results（no blood transfusion within 14 days）：

   1. Hemoglobin（HB）≥90g/L；
   2. Absolute neutrophils count（ANC）≥1.5×109/L；
   3. Blood platelets（PLT）≥80×109/L
2. Biochemical tests results defined as follows：

   1. Total bilirubin（TBIL）≤1.5 times the upper limit of normal (ULN) ；
   2. Alanine aminotransferase（ALT）and aspartate aminotransgerase AST≤2.5ULN，liver metastases，if any，ALT和AST≤5ULN；
   3. Creatinine（Cr）≤1.5ULN or Creatinine Clearance rate (CCr)≥60 ml/min；
3. Doppler ultrasound assessment：left ventricular ejection fraction (LVEF) ≥the lower limit of normal value(50%).

Exclusion Criteria:

1. Small cell lung cancer(including patients with mixed small cell lung cancer and non-small cell lung cancer) or central squamous cell carcinoma with cavity
2. Mutation status are unknown
3. Previously (within 5 years) or presently suffering from other malignancies,
4. Symptomatic or uncontrolled brain metastases
5. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months or serious cardiac arrhythmia requiring medication
6. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications
7. Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation, or prior surgical procedures affecting absorption
8. Pregnancy or lactation
9. Previously treated including treated with traditional Chinese medicine
10. Patients who are allergic to any of the agent or any ingredient -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety will be assessed according to common terminology criteria for adverse events version 4.0 (CTC AE 4.0) | from initiation of treatment to 90 days after the treatment finished
ORR | at the time of 8 weeks (2 cycles after treatment)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1). The percentage of patients who achieved CR and PR was defined as objective response rate (ORR)

SECONDARY OUTCOMES:
DCR | at the time of 8 weeks (2 cycles after treatment)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1) and the percentage of patients who achieved CR, PR and SD was defined as disease control rate (DCR).
PFS | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause.
OS | From date of treatment until the date of death from any cause, assessed up to 50 months
  OS is calculated from diagnosis to death or last follow-up time.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The data used or analyzed during the current study are available from the principle investigator on reasonable request after 6 months of the project is finished.

REFERENCES:
- [Derived] Chu T, Zhong R, Zhong H, Zhang B, Zhang W, Shi C, Qian J, Zhang Y, Chang Q, Zhang X, Dong Y, Teng J, Gao Z, Qiang H, Nie W, Zhao Y, Han Y, Chen Y, Han B. Phase 1b Study of Sintilimab Plus Anlotinib as First-line Therapy in Patients With Advanced NSCLC. J Thorac Oncol. 2021 Apr;16(4):643-652. doi: 10.1016/j.jtho.2020.11.026. Epub 2021 Jan 29. PMID 33524601